CLINICAL TRIAL: NCT02256826
Title: Study of Pharmacokinetic Interaction Between Kaletra® (LPV/r) and BILR 355 BS Plus Ritonavir
Brief Title: Study of Pharmacokinetic Interaction Between Kaletra® (LPV/r) and BILR 355 BS Plus Ritonavir in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1188.8
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Ritonavir; lopinavir-ritonavir drug combination

ARMS (2):
- Group A (Experimental)
  Interventions: Drug: BILR 355 BS; Drug: Ritonavir (RTV); Drug: Kaletra®
- Group B (Experimental)
  Interventions: Drug: BILR 355 BS; Drug: Ritonavir (RTV)

INTERVENTIONS:
Drug: BILR 355 BS
Drug: Ritonavir (RTV) — NORVIR®
Drug: Kaletra® — (lopinavir (LPV) and ritonavir (RTV))
  Arms: Group A

SUMMARY:
To determine the pharmacokinetic effect of BILR 355 BS on Kaletra® and of Kaletra® on BILR 355 BS

ELIGIBILITY:
Inclusion Criteria:

1. Males or females who meet the inclusion/exclusion criteria; females must not be pregnant or nursing, and agree to use a double-barrier method of birth control (condoms or diaphragm plus spermicide) throughout the trial (alone or in addition to other methods of birth control such as oral contraceptives)
2. Age ≥18 and <60 years
3. BMI ≥18.5 and BMI ≤29.9 kg/m2
4. Ability to give signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local regulations

Exclusion Criteria:

1. Current (symptomatic within the last 30 days) and medically relevant gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
2. Surgery of gastrointestinal tract (except appendectomy)
3. Currently active (symptomatic within the last 30 days) diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
4. History of relevant orthostatic hypotension, fainting spells or blackouts
5. History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
6. Intake of drugs with a long half-life (>24 hours) within one month prior to administration of study drug or during the trial (review with clinical monitor if questionable)
7. Use of drugs within 10 days prior to administration or during the trial, which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation (review with clinical monitor if questionable)
8. Participation in another trial with an investigational drug within one month prior to administration or during the trial
9. Current smoker
10. Alcohol (more than 60 g/day) or drug abuse (positive urine test for illicit prescription or non-prescription drugs or drugs of abuse)
11. Recent blood donation (more than 100 mL within 4 weeks prior to administration or during the trial)
12. Excessive physical activities (within 1 week prior to study drug administration or during the trial)
13. Any laboratory value outside the normal reference range that is of clinical relevance at screening, according to the judgment of the investigator
14. Inability to comply with dietary regimen required by the protocol
15. Chronic or relevant acute infections
16. Infected with hepatitis B or hepatitis C viruses (defined as either being hepatitis B surface antigen, or hepatitis C antibody positive)
17. HIV-1 infected as defined by a positive HIV ELISA test

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2005-04; Primary Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over one dosing interval (12 hours) at steady state (AUC0-12h,ss) | Up to 12 h after the last drug administration of BILR 355
Maximum measured concentration of the analyte in plasma at steady state over a dosing interval τ (Cmax,ss) | Up to 96 h after the last drug administration of BILR 355

SECONDARY OUTCOMES:
Apparent clearance of the analyte in plasma following extravascular administration at steady state (CL/F,ss) | Up to 96 h after the last drug administration of BILR 355
Time from dosing to the maximum concentration of the analyte in plasma at steady state (tmax,ss) | Up to 96 h after the last drug administration of BILR 355
Terminal half-life of the analyte in plasma at steady state (t1/2,ss) | Up to 96 h after the last drug administration of BILR 355
Apparent volume of distribution during the terminal phase λz at steady state following an extravascular dose (Vz/F,ss) | Up to 96 h after the last drug administration of BILR 355
Area under the plasma concentration time curve (0-12 hours) (AUC0-12h) for RTV | Up to 12 h after RTV administration
Maximum measured concentration of the analyte in plasma at steady state (Cmax,ss) for RTV | Up to 96 h after the last drug administration of BILR 355
Measured concentration of the analyte in plasma 12 hours post last dose at steady state (Cp12h,ss) | Up to 12 h after the last drug administration of BILR 355
Number of participants with Adverse Events | Up to day 35 after first drug administration
Number of participants with abnormal changes in clinical laboratory parameters | Up to day 35 after first drug administration
Number of participants with abnormal findings in physical examination | Up to day 35 after first drug administration
Number of participants with clinically significant changes in vital signs | Up to day 35 after first drug administration